CLINICAL TRIAL: NCT05568459
Title: A Prospective Study to Evaluate Disease Characteristics in Hemophilia B Participants Receiving Prophylaxis With Standard of Care FIX Replacement Therapy
Brief Title: A Trial That Evaluates Disease Characteristics in Hemophilia B Adult Male Participants Receiving Prophylaxis With Standard of Care Factor IX Protein (FIX) Replacement Therapy
Acronym: Honey-B
Status: Active, not recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R0000-HEMB-2187
Record Dates: First submitted 2022-09-23; First posted 2022-10-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hemophilia B
Keywords: FIX replacement therapy
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Male participants with hemophilia B on current FIX Replacement Therapy prophylaxis or a documented genotype known to produce severe hemophilia B
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — No study treatment will be administered in this study.

SUMMARY:
This study is focused on males who have Hemophilia B and who need regular preventive treatment with factor IX protein (FIX) replacement therapy to prevent and also to control their bleeding events. The aim of the study is to gather at least 6 months of information on bleeding events for each individual participant while they continue to use their usual FIX replacement therapy. There is no experimental treatment being tested in this study. The study is informational, and part of a larger program to understand and treat Hemophilia B with a potential experimental new therapy in the future. There is no obligation to agree to taking part in this future study.

The study is looking to answer several other research questions to help understand each participant's individual disease characteristics, including:

* How often to use FIX replacement therapy, both on a regular basis (prophylaxis) and as needed to treat bleeding events
* Measurement of FIX activity (factor IX is a clotting factor) by different laboratories using different types of tests in Hemophilia B participants
* Possible complications from the FIX replacement therapy the patient receives (usual standard of care will continue to be used)
* How quality of life is affected by Hemophilia B
* How joint health is affected by Hemophilia B
* How often the participant visits the emergency room, urgent care center, physician's office, hospital, or has a telemedicine visit as a result of bleeding events
* Whether the body makes antibodies (a protein produced by the body's immune system) against the FIX replacement therapy you receive, which could make the drug less effective or could lead to side effects

ELIGIBILITY:
Key Inclusion Criteria:

1. Previous experience with FIX therapy (≥50 documented exposure days to a FIX protein product such as recombinant, plasma-derived or extended half-life FIX product) with a current stable prophylaxis regimen for >2 months prior to enrollment and intention to use FIX replacement therapy for the duration of the study
2. No known hypersensitivity to FIX replacement product
3. Willing to be contacted about a potential future clustered regularly interspaced short palindromic repeats (CRISPR)-based Factor 9 (F9) gene insertion clinical trial in which they may have the opportunity to screen for enrollment

Key Exclusion Criteria:

1. History of any coagulation disorder; requires anticoagulant therapy
2. Lack of adherence with documentation of bleeds and/or prophylaxis replacement therapy administration in the opinion of the investigator, based on medical history
3. History of FIX inhibitor (clinical or laboratory-based assessment) on 2 or more occasions, as defined in the protocol
4. Bethesda inhibitor titer greater than the upper limit of normal (ULN) at screening
5. Any detectable pre-existing antibodies to the Adeno-associated virus serotype 8 (AAV8) capsid; as measured by an assay at prescreening, as defined in the protocol
6. Is positive for hepatitis B or C at screening, as defined in protocol
7. If any of the following pre-existing diagnoses are documented:

   * Cholestatic liver disease
   * Liver cirrhosis
   * Portal hypertension; or
   * Splenomegaly; or
   * Hepatic encephalopathy
8. History of arterial or venous thrombo-embolic events, as defined in the protocol
9. History of clinically significant cardiovascular, respiratory, hepatic, renal (including nephrotic syndrome), gastrointestinal (including protein-losing enteropathy), endocrine, hematological (including thrombophilia), psychiatric, or neurological disease, as assessed by the investigator that may confound the results of the study or poses an additional risk to the participant by study participation
10. Previously received of any AAV-gene based therapy with a marketed gene therapy or in a clinical trial or intent to receive approved or investigational AAV-gene based therapy during the study period

NOTE: Other Inclusion/Exclusion Protocol Defined Criteria Apply

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male with moderately severe to severe Hemophilia B with medical history of FIX functional activity/ FIX:C (≤2% or <0.02 IU/mL) or a documented genotype known to produce severe hemophilia B
Study Population: Male patients with Hemophilia B with a history of FIX:C ≤2% or a documented genotype known to produce severe hemophilia B on current FIX Replacement Therapy prophylaxis
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
Annualized bleeding rate (ABR) | At least 26 Weeks Up to 96 weeks

SECONDARY OUTCOMES:
Annualized utilization (IU/kg) of FIX replacement therapy | Up to 96 Weeks
FIX functional (coagulant) activity (FIX:C) in participants on prophylaxis FIX replacement therapy | Through the end of the study, approximately 96 Weeks
  FIX:C includes pre-dose and average activity
Difference of FIX:C in participants on prophylaxis FIX replacement therapy by one-stage and chromogenic assays | Through the end of the study, approximately 96 weeks
Difference of FIX:C between one-stage assay and chromogenic substrate assay by laboratory in participants on prophylaxis FIX replacement therapy | Through the end of the study, approximately 96 weeks
Difference of FIX:C between laboratories by assay (one-stage assay and chromogenic substrate assay) in participants on prophylaxis FIX replacement therapy | Through the end of the study, approximately 96 weeks
Incidence of adverse event (AEs) | Through the end of the study, approximately 96 Weeks
Severity of AEs | Through the end of the study, approximately 96 Weeks
Hemophilia Quality of Life (Haemo-Qol-A) total and individual domain scores | Up to 96 Weeks
  The Haemo-QoL-A is a self-reported Hemophilia-specific health-related quality of life questionnaire which consists of 41 questions covering 6 domains (Physical Functioning, Role Functioning, Worry, Consequences of Bleeding, Emotional Impact, and Treatment Concerns). Items are answered on a 6-point Likert-type scale, ranging from 0 (None of the time) to 5 (All of the time). Higher scores mean better health-related quality of life or less impairment.
Hemophilia Activities List (HAL) total and individual scores | Up to 96 Weeks
  HAL measures of the impact of Hemophilia on functional abilities in adults. The questionnaire consists of 42 items across 7 domains. Each item is rated on a scale of 1 (Impossible) to 6 (Never). Higher scores represent lower levels of activity limitations.
European Quality of Life 5 Dimensions 3-levels (EQ-5D-3L) score | Up to 96 Weeks
  EQ-5D-3L health questionnaire is a participant/relative answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. the status of each dimension had 3 possible responses (1 =no problem, 2 some problem 3 =severe problems) in the relevant health dimension. Higher score indicated a worsening health condition.
Hemophilia Joint Health Score (HJHS) total and individual scores per joint | Up to 96 Weeks
  The examination involves a physical assessment of elbow, knee, and ankle joints. Individual joints are scored based on duration and presence of swelling, joint pain, flexibility, muscle atrophy, strength, and overall gait. The HJHS is a validated 11-item scoring tool based on radiologic and clinical evaluation, sensitive to detect early signs and minor changes. HJHS ranges from 0 to 124. Higher values in the HJHS represent worse situation for the participant.
Annualized medically attended visit (MAV) rate for any reason | Up to 96 Weeks
  The annual rate of MAVs including emergency room (ER) visits, urgent care center visits, physician's office visits, telemedicine visits, or hospitalizations related to bleeds treated on-demand with FIX replacement therapy
Detection of antibodies to adeno-associated virus (AAV) capsid proteins | Up to 96 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (17):
- United States (9):
  - University of Colorado Hemophilia and Thrombosis Center, Aurora, Colorado
  - Yale HTC, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Texas Health Science Center at Houston, Houston, Texas
- Canada (2):
  - McMaster University Medical Centre - Hamilton Health Sciences, Hamilton, Ontario
  - Mcgill University Health Center (MUHC), Montreal, Quebec
- Germany (3):
  - University Hospital of Regensburg, Regensburg, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet Frankfurt, Frankfurt
  - University Hospital Hamburg Eppendorf, Hamburg
- United Kingdom (3):
  - Southampton General Hospital, Southampton, Hampshire
  - Barts Health NHS Trust, Royal London Hospital, London
  - St. Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/